CLINICAL TRIAL: NCT01559818
Title: An Open Label Long Term Follow up Study for Patients With Melanoma Who Were Previously Enrolled in the Phase I Study IMM-101-001
Brief Title: A Long Term Follow up Study for Patients Who Previously Took Part in the Phase I Study IMM-101-001
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor considered no further meaningful data was being collected, nor were likely to be collected in the future.
Sponsor: Immodulon Therapeutics Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMM-101-008
Record Dates: First submitted 2012-03-19; First posted 2012-03-21 (Estimated); Results first posted 2023-05-24 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2022-07

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma | interventions — IMM-101

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IMM-101 (Experimental): IMM-101 1.0 mg administered intradermally
  Interventions: Biological: IMM-101

INTERVENTIONS:
Biological: IMM-101 — IMM-101 10mg/mL, a suspension of heat-killed whole cell M. obuense in borate-buffered saline.
  Other Names: Heat-killed whole cell M. obuense

SUMMARY:
Patients who were previously enrolled in Study IMM-101-001 and who provided informed consent were eligible to participate in this study.

Once eligibility was confirmed, a full medical history covering the period from completion of Study IMM-101-001 to date was taken.

The treatment regimen with IMM-101 was one dose given every 4 weeks or as close to this interval as permitted due to practical or logistic considerations. The dose interval could be modified at the discretion of the Investigator provided the minimum period between doses was no less than 14 days.

The overall objective was to determine the long term safety profile of IMM-101 administered intradermally for extended use.

DETAILED DESCRIPTION:
This was an open-label long term follow up study. The study consisted of two phases:

1. Screening and enrolment Patients, who provided informed consent participated in a screening period of up to 28 days to establish eligibility. Once eligibility was confirmed a full disease and treatment history covering the period from their completion of Study IMM-101-001 to date was taken.
2. Treatment Patients could receive ongoing treatment every 4 weeks or as close to this interval as permitted due to practical or logistic considerations until death or withdrawal, unless such therapy was contraindicated, the patient did not wish to continue or the study was terminated by the Sponsor. At no point could the elapsed period between IMM-101 doses be less than 14 days.

Patients could choose to withdraw from the study at any time and for any reason. IMM-101 could be stopped or the dosing regimen reduced if felt to be necessary by the Investigator and/or patient (e.g., intolerable injection site reactions).

In the event of an injection site reaction of Grade 3 and above, and/or if significant ulceration, tenderness or lymphadenopathy was observed, at the discretion of the Investigator, patients could be administered a half dose of the study drug (i.e., a single 0.05 mL intradermal injection of IMM-101) or the timing of the injection could be delayed. If the dosing interval was increased, the patient still attended the study site for safety assessments preferably every 3 months but, if this was not possible, every 6 months at a minimum. The blood sample for exploratory analysis continued to be taken every 6 months.

Any change in the dose of study drug administered or the frequency of dose administration was recorded in the patient's case report form (CRF). In the case of withdrawal, separate consent was sought to allow the continued collection on patient status.

ELIGIBILITY:
Inclusion Criteria:

* Patient was previously enrolled in Study IMM-101-001
* Patient gave consent to make their disease and treatment history for the intervening period between their completion of Study IMM-101-001 and enrollment in this study available to the Sponsor
* Patient gave signed informed consent for participation in the study

Exclusion Criteria:

* Female patient of child-bearing potential who was not, in the opinion of the Investigator, using an approved method of birth control (e.g., physical barrier [patient and partner], contraceptive pill or patch, spermicide and barrier, or intrauterine device [IUD]).

Those patients that utilised hormonal contraceptives must have used the same method for at least three months before additional barrier contraception (as described above) was discontinued from being used concomitantly with the hormonal contraception.

* Patient of non-child-bearing potential were defined as having 12 month amenorrhoea or were surgically sterile.
* Female patient who was pregnant, breast feeding or planning a pregnancy during the course of the study. A pre-treatment urine pregnancy test measuring human chorionic gonadotrophin (hCG) must be negative.
* Patient was unable or unwilling to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Fusi, Dr, Principal Investigator — St George's, University of London
Locations (1):
- St Georges University of London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IMM-101
Started | 10
Completed | 3
Not Completed | 7
Not completed — Physician Decision | 1
Not completed — Pregnancy | 1
Not completed — Study terminated by Sponsor | 4
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: All enrolled patients
Groups:
- IMM-101: IMM-101 1.0 mg I.D.
  IMM-101: IMM-101 10mg/mL, a suspension of heat-killed whole cell M. obuense in borate-buffered saline.
Arm/Group | IMM-101
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants] — This study and the preceding IMM-101-001 study were conducted in the United Kingdom only
  Participants
    United Kingdom | 10

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events With a Causal Relationship to IMM-101
Description: Adverse events measured throughout the study and assessed for severity using NCI CTCAE and causality to measure the profile and number of local and systemic toxicities. Treatment related Adverse Events were defined as being definitely, probably or possibly related to IMM-101 or with an unknown relationship.
Time Frame: From the time of signing informed consent until 30 days after the end of study or withdrawal, a median of 4.4 years (range 1.2 to 6.7).
Population: Safety population = all enrolled patients
Measure: Number; unit: Events
Arm/Group | IMM-101
Number analyzed (Participants) | 10
Events | 27

2. Primary Outcome: Treatment Emergent Adverse Events of NCI CTCAE ≥Grade 3
Description: Adverse events measured throughout the study and assessed for severity using NCI CTCAE and causality to measure the profile and number of local and systemic toxicities
Time Frame: as for outcome 1
Population: Safety population = all enrolled patients
Measure: Number; unit: Events
Arm/Group | IMM-101
Number analyzed (Participants) | 10
Events | 16

3. Primary Outcome: Treatment Emergent Serious Adverse Events
Description: Adverse events measured throughout the study and assessed for severity using NCI CTCAE and causality to measure the profile and number of local and systemic toxicities.
  There were no IMM-101 related serious adverse events reported during the study.
Time Frame: as for outcome 1
Population: Safety population = all enrolled patients
Measure: Number; unit: Events
Arm/Group | IMM-101
Number analyzed (Participants) | 10
Events | 3

4. Secondary Outcome: Survival
Description: Overall survival
Time Frame: Overall survival was defined as the time from enrolment until date of death for up to 81 months. Patients still alive after 81 months were censored at withdrawal from the study or at last known date alive if later.
Population: There was only one analysis population in the study. Safety, tolerability and efficacy endpoints were summarised using the safety population, defined as all patients who received at least one dose of the study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | IMM-101
Number analyzed (Participants) | 10
Participants
  Died | 3
  Censored | 1
  Alive | 6

5. Secondary Outcome: Incidence of Change in Metastatic Disease
Description: The protocol required any change in metastatic disease to be documented where possible. However, given this was a real-life long-term follow-up study, CT or MRI scans were not mandated as part of the protocol and were only performed as clinically indicated. Very few scans were performed during the course of the study (0 to nine events per patient). Given the fact patients could receive anti-cancer therapy on study, disease status fluctuated throughout the study (better, worse, no change). This coupled with the sparsity of CT or MRI scan data collected on a per patient basis resulted in only Best Overall Response being described.
Time Frame: From Informed Consent to death or withdrawal (median 4.4 years, range 1.2 - 6.7)
Population: All enrolled patients
Measure: Number; unit: participants
Arm/Group | IMM-101
Number analyzed (Participants) | 10
participants
  Best Overall Response = Not known | 1
  Best overall response = Improved | 4
  Best Overall Response = No Change / Stable Disease | 4
  Best Overall Response = Disease worsening | 1

6. Other Pre Specified Outcome: Translational Research
Description: Blood samples were collected and sera prepared for analysis of immunological markers and mediators.
  Exploratory endpoints may include a change in one or more markers of immune status based on cellular involvement, function or cytokine/immune mediator production such as, for example, cytokines and antibodies, or any other clinically or immunologically relevant assays.
Time Frame: From baseline to death or withdrawal
Population: Extensive translational research on serum samples from other studies with IMM-101 failed to identify any clinically significant impact on relevant immunological markers or mediators. Therefore no analysis was perform on the samples from this study.
Arm/Group | IMM-101
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of informed consent until study completion (median 4.4 years, range 1.2 - 6.7)
Description: Adverse events (including those reported spontaneously by the patient, observed by the Investigator or elicited using non-leading questions) were collected from the time of signing informed consent until 30 days after the end of study or withdrawal.
  Adverse event information could be obtained during study visits or by telephone contact with the patient between visits.
Groups:
- IMM-101: IMM-101 1.0 mg I.D.
Arm/Group | IMM-101
All-Cause Mortality (participants affected / at risk) | 4/10
Serious Adverse Events (participants affected / at risk) | 2/10
Other Adverse Events (participants affected / at risk) | 7/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMM-101 (N=10)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMM-101 (N=10)
Injection site reaction (General disorders) | 6 (12)
Injection site pain (General disorders) | 1 (1)
Influenza like illness (General disorders) | 1 (1)
Injection site ulcer (General disorders) | 1 (3)
Fatigue (General disorders) | 1 (1)
Injection site erythema (General disorders) | 1 (1)
Injection site infection (General disorders) | 1 (1)
Injection site necrosis (General disorders) | 1 (1)
Injection site swelling (General disorders) | 1 (1)
Peripheral swelling (General disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Night sweats (Nervous system disorders) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (2)

LIMITATIONS AND CAVEATS:
The median survival time was not calculable as less than 50% patients died. No inferences can be made from the rate of survival due to the small sample size.

Given the fact patients could receive anti-cancer therapy on study, disease status fluctuated throughout the study (better, worse, no change). This coupled with the sparsity of CT or MRI scan data collected on a per patient basis resulted in only Best Overall Response being described.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-06-05): https://cdn.clinicaltrials.gov/large-docs/18/NCT01559818/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-10): https://cdn.clinicaltrials.gov/large-docs/18/NCT01559818/SAP_001.pdf